CLINICAL TRIAL: NCT00920803
Title: A Phase 1, Double-Blind, Randomized Clinical Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of SRT501 in Subjects With Colorectal Cancer and Hepatic Metastases
Brief Title: A Clinical Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of SRT501 in Subjects With Colorectal Cancer and Hepatic Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 113221
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Neoplasms, Colorectal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5g SRT501 (Active Comparator): 5.0 g of SRT501 will be administered once daily as an oral reconstituted powder, for 14 days at the same time each day. On Days 1 and 2, SRT501 will be administered approximately 15-30 minutes following the consumption of a standardized breakfast. On all other days, SRT501 will be administered approximately 15-30 minutes following the consumption of the evening meal. Following the course of SRT501 administration, subjects will undergo scheduled surgical removal of their metastatic liver disease as well as non-diseased tissue. Due to scheduling and surgical availability, subjects can receive SRT501 for a minimum of 10 days and a maximum of 21 days.
  Interventions: Drug: SRT501
- Placebo (Placebo Comparator): Placebo will be administered once daily as an oral reconstituted powder, for 14 days at the same time each day. On Days 1 and 2, placebo will be administered approximately 15-30 minutes following the consumption of a standardized breakfast to allow for PK sample collection. On all other days, placebo will be administered approximately 15-30 minutes following the consumption of the evening meal. Following the course of placebo administration, subjects will undergo scheduled surgical removal of their metastatic liver disease as well as non-diseased tissue. Due to scheduling and surgical availability, subjects can receive placebo for a minimum of 10 days and a maximum of 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo will be supplied in clinical kits as a powder which will be reconstituted with vehicle and water into a liquid suspension. Placebo must be used immediately following mixing. Placebo will be administered orally, once daily for 14 days.
  Arms: Placebo
Drug: SRT501 — SRT501 will be supplied in clinical kits as a powder which will be reconstituted with vehicle and water into a liquid suspension. The final drug product must be used immediately following mixing. SRT501 will be administered orally, once daily for 14 days.
  Arms: 5g SRT501

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of SRT501 (5.0 g) in subjects with colorectal cancer and hepatic metastases when administered once daily for 14 days.

The purpose is to also characterize the pharmacokinetic profile of SRT501 (5.0 g) by assessing levels of SRT501 and metabolites in blood, urine, bile and normal and malignant metastatic tissues in subjects with colorectal cancer and hepatic metastases when administered once daily for 14 days.

The secondary purpose is to examine the pharmacodynamics of SRT501 activity in both normal and malignant tissue samples, including blood and/or bodily fluids.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, inpatient/outpatient study to assess the safety, pharmacokinetics, and pharmacodynamics of SRT501 in subjects diagnosed with colorectal cancer and hepatic metastases. Fifteen subjects aged 18 years of age and older who fulfill the inclusion/exclusion criteria, will be enrolled in this study. Ten subjects, if eligible, will be randomized to receive SRT501 and 5 subjects, if eligible, will be randomized to receive placebo. Subjects will sign the informed consent form prior to any study-related procedures. If eligible, subjects will consent to receive 5.0 g of SRT501 or placebo, to be administered once daily as an oral reconstituted powder, for 14 days at the same time each day. On Days 1 and 2, SRT501 or placebo will be administered approximately 15-30 minutes following the consumption of a standardized breakfast to allow for PK sample collection. On all other days, SRT501 or placebo will be administered approximately 15-30 minutes following the consumption of the evening meal. Following the course of SRT501 or placebo administration, subjects will undergo scheduled surgical removal of their metastatic liver disease as well as non-diseased tissue and these samples will be evaluated for SRT501 concentrations and pharmacodynamic markers of neoplastic activity (such as cell differentiation, apoptosis, proliferation, etc.). Due to scheduling and surgical availability, subjects can receive SRT501 or placebo for a minimum of 10 days and a maximum of 21 days. If diseased colon tissue is also scheduled to be removed during resection, both diseased and normal colon tissue will also be collected for analysis. Participants will be required to return to the study center on Day 2 for a 24-hour PK sample and the evening prior to their scheduled surgical resection as well as per the Institution's standards of care for recovery following the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female greater than 18 years of age.
* Have histologically or cytologically confirmed and diagnosed colorectal cancer with hepatic metastases.
* Have not received chemotherapy or anti-neoplastic therapy for a malignancy within six weeks of first dose of SRT501 or placebo.
* Have a life expectancy of greater than 3 months.
* Voluntarily sign an Ethics Committee (EC)-approved informed consent form (ICF) to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.
* Be deemed, in the Investigator's opinion, to be able to physically comply with SRT501 dosing.
* Be amenable to surgical resection of the hepatic metastases.
* Be clear of any history of HIV 1 and 2 and hepatitis B and C.
* Have a normal 12-lead ECG or an ECG with abnormality considered to be clinically insignificant.
* Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
* Female subject is either post-menopausal, surgically sterilized or be a woman of child bearing potential (WCBP) who has documented use of clinically prescribed hormonal contraceptives use consistently for three months prior to study entry. Females of child bearing potential, as well as their partners, must also use appropriate double-barrier birth control while participating in the study and for 28 days following the last dose of study drug. If a woman of child bearing potential has a surgically sterile partner, then that female is permitted to enroll if double-barrier birth control is practiced.

Exclusion Criteria:

* Subject has a history / evidence of allergy or hypersensitivity to resveratrol.
* Subject has had a major illness (other than colorectal cancer) in the past three months or any significant ongoing chronic medical illness that the Investigator would deem unfavorable for enrollment.
* Subject has inadequate organ function at the Screening visit as defined by the following laboratory values:

  * Platelet count ≤100,000 x 10^9/L
  * Hemoglobin ≤10.0 g/dL
  * Subjects with lower hemoglobin may be included at the Investigator's discretion if the cause of anemia is due to bleeding from their tumor and post transfusion hemoglobin ≥10g/dL prior to dosing.
  * Absolute neutrophil count (ANC) ≤1500 x 10^6/L
  * Aspartate transaminase (AST) ≥2.5 x the upper limit of the normal range (ULN)
  * Alanine transaminase (ALT) ≥2.5 x ULN
  * Creatinine ≥ 140 umol/L
  * Albumin ≤3 g/dL
* Subject has a history of or current gastro-intestinal diseases influencing drug absorption, with the exception of an appendectomy and/or colorectal cancer.
* Subject has liver impairment as indicated by total bilirubin ≥2 x ULN, unless clearly related to the disease (ie, biliary occlusion due to tumor compression or confirmed Gilbert's Disease as documented by the Investigator).
* Subject had a myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Excessive alcohol intake (more than UK recommended limit - 28 or 21 units per week for men or women respectively).
* Subject has uncontrolled brain metastases or central nervous system disease.
* Subject has participated in a clinical trial within the past three months.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-hCG pregnancy test result obtained during the Screening period. Pregnancy testing is not required for post-menopausal or surgically sterilized women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08-19 (Actual); Primary Completion 2009-11-11 (Actual); Study Completion 2009-11-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of SRT501 when administered once daily for 14 days. | Safety will be continually assessed while subjects are on study.
To characterize the pharmacokinetic profile of SRT501 in blood and normal and malignant metastatic tissues when administered once daily for 14 days. | Pharmacokinetic samples will be obtained on Days 1, 2, 14, and 15.

SECONDARY OUTCOMES:
To examine the pharmacodynamics of SRT501 activity in both normal and malignant tissue samples and blood. | Pharmacodynamic samples will be collected on Days 14 and 15 and will be analyzed at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Howells LM, Berry DP, Elliott PJ, Jacobson EW, Hoffmann E, Hegarty B, Brown K, Steward WP, Gescher AJ. Phase I randomized, double-blind pilot study of micronized resveratrol (SRT501) in patients with hepatic metastases--safety, pharmacokinetics, and pharmacodynamics. Cancer Prev Res (Phila). 2011 Sep;4(9):1419-25. doi: 10.1158/1940-6207.CAPR-11-0148. Epub 2011 Jun 16. PMID 21680702
- See also: Results for study 113221 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113221?search=study&search_terms=113221#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register